CLINICAL TRIAL: NCT07275190
Title: The Use of Machine Learning Techniques for the Differential Diagnosis Between Eosinophilic Granulomatosis With Polyangiitis and Hypereosinophilic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carlomaurizio Montecucco, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AI_EH_resub
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: EGPA - Eosinophilic Granulomatosis With Polyangiitis; HES - Hypereosinophilic Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome; Hypereosinophilic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood draw for the laboratory assessment — Blood draw for the laboratory assessment

SUMMARY:
The purpose of this study is to collect clinical, laboratory, and instrumental data from patients with eosinophilic granulomatosis with polyangiitis or hypereosinophilic syndrome, which will then be analyzed using artificial intelligence techniques with the aim of identifying characteristics that differentiate the two diseases and can predict the response to the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or over
2. A diagnosis of EGPA or HES
3. Willing and able to give informed written consent, or willing to give permission for a nominated friend or relative to provide written informed assent if they are unable to do so because of physical disabilities

Exclusion Criteria:

1. Lack of a confirmed diagnosis of EGPA or HES.
2. Other causes of eosinophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
characteristics that are different between HES and EGPA | 18months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Reumatologia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No